CLINICAL TRIAL: NCT04712747
Title: Adaptive Optics (AO) Analysis of Retinal Arteries in Patients With Recent Stroke (STROKAO)
Acronym: STROKAO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2020_28
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Adaptive optics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases - patients with stroke: Ophthalmological examinations : At the inclusion visit and 3 months after their stroke Blood pressure measurement at rest : At the inclusion visit
  Interventions: Procedure: Ophthalmological examinations; Procedure: Blood pressure measurement at rest
- Controls - Individuals with no history of stroke: Ophthalmological examinations : At the inclusion visit Blood pressure measurement at rest : At the inclusion visit
  Interventions: Procedure: Ophthalmological examinations; Procedure: Blood pressure measurement at rest

INTERVENTIONS:
Procedure: Ophthalmological examinations — * OCT (Optical Coherence Tomography): posterior pole OCT B scan , optic nerve and posterior pole OCT Angiography
  * Adaptive optics (AO) : Image acquisition on the vessels at the exit of the optic nerve before the first upper temporal bifurcation OD or OG and evaluation of the photoreceptor mosaic. Adaptive optics may require dilatation of the pupil with a drop of tropicamide in the eye examined a few minutes before the examination.
  * Color retinophotography
  * Measurement of intraocular pressure
  Patients with stroke : At the inclusion visit and 3 months after their stroke Control group : At the inclusion visit.
Procedure: Blood pressure measurement at rest — At the inclusion visit

SUMMARY:
The eye has long been recognized as a window to pathological processes occurring in the brain. By imaging the vascular system of the retina scientific understanding and clinical practice have been improved for a wide range of pathologies from diabetes to stroke and dementia.

Adaptive optics (AO) reveals retinal details that remain invisible with other current imaging techniques. Indeed, vessels can be perfectly visualized, making it possible to detect wall irregularities, accurately measure their different structures and monitor their evolution under treatment if necessary.

In AO, studies on retinal vessels involve the calculation of wall thickness (WT), outer diameter (OD), inner diameter (ID), wall cross-sectional area (WCSA) and wall to lumen ratio (WLR). An increase in WLR > 0.31 is characteristic of hypertensive microangiopathy and predictive of cardiovascular and brain damage. This accurate assessment of microvascular structure may even be required in the near future in all patients with arterial hypertension. For vessels > 300 microns in diameter, the increase in vessel wall thickness occurs without changing the ID, a process known as external hypertrophic remodeling. For small arteries < 300 microns, remodeling occurs differently. The total volume of the vessel wall remains constant, but the OD and ID each decrease, a process known as inward eutrophic remodeling.

The objective of this study is to describe the parameters measured in AO in patients in the acute phase of a stroke and then at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* For the patients with stroke: Inpatients with confirmed stroke (clinical and imaging) for less than 10 days
* For the controls: Individuals presenting at the Rothschild Foundation Hospital with no history of stroke who are matched to cases already included in the matching criteria: Age ± 5 years, Gender, high blood pressure (no history, untreated, treated) Diabetes (Yes, No), Body Mass Index (BMI < 25, 25 ≥ BMI < 30, BMI ≥ 30)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Insufficient state of consciousness or physical condition to perform the adaptive optics examination
* For the patients with stroke: Hemorrhagic post-traumatic hematoma stroke type, or symptomatic stroke of a brain tumour or an arteriovenous malformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients with confirmed stroke for less than 10 days and controls (Individuals presenting at the Rothschild Foundation Hospital with no history of stroke)
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Wall thickness (WT) in adaptive optics | At the inclusion visit (less than 10 days after the stroke for the patients with stroke)
  Measured in µm², Comparison between groups : hemorrhagic strokes, ischemic strokes, controls
Wall cross-sectional area (WCSA) in adaptive optics | At the inclusion visit (less than 10 days after the stroke for the patients with stroke)
  Measured in µm², Comparison between groups : hemorrhagic strokes, ischemic strokes, controls
Wall to lumen ratio (WLR) in adaptive optics | At the inclusion visit (less than 10 days after the stroke for the patients with stroke)
  Comparison between groups : hemorrhagic strokes, ischemic strokes, controls

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France